CLINICAL TRIAL: NCT00666926
Title: A Phase 1, Open-Label, Dose Escalation Study To Evaluate Safety, Pharmacokinetics And Pharmacodynamics Of PF-00562271 In Patients With Advanced Non-Hematologic Malignancies
Brief Title: Study Of PF-00562271, Including Patients With Pancreatic, Head And Neck, Prostatic Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A8031001
Record Dates: First submitted 2008-03-26; First posted 2008-04-25 (Estimated); Results first posted 2012-06-14 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Head and Neck Neoplasm; Prostatic Neoplasm; Pancreatic Neoplasm
Keywords: Pancreatic Neoplasm; Head and Neck neoplasm; Prostatic neoplasms; Focal Adhesion Kinase; Phase 1; Pharmacodynamics; FDG-PET
MeSH Terms: conditions — Head and Neck Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms | interventions — PF-00562271

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: PF00562271
- 2 (Experimental)
  Interventions: Drug: PF00562271
- 3 (Experimental)
  Interventions: Drug: PF00562271
- 4 (Experimental)
  Interventions: Drug: PF00562271

INTERVENTIONS:
Drug: PF00562271 — 125 mg twice daily [BID] with food, tablet
  Arms: 1
Drug: PF00562271 — 125 mg BID with food, tablet
  Arms: 2
Drug: PF00562271 — 125 mg BID with food, tablet
  Arms: 3
Drug: PF00562271 — 125 mg BID with food, tablet
  Arms: 4

SUMMARY:
Phase 1 safety, pharmacokinetics, and pharmacodynamics trial of the focal adhesion kinase (FAK) inhibitor PF-00562271 in patients with positive Positron Emission Tomography [PET] scans due to advanced non-hematologic malignancies, including pancreatic, head and neck, and prostatic neoplasms, and patients with other malignancies appropriate for serial biopsy. Screening consists of a Fluorodeoxyglucose Positron Emission Tomography [FDG-PET] and tumor imaging, medical history, physical examination, Eastern Cooperative Oncology Group [ECOG] performance status, blood draws, a pregnancy test for female patients of childbearing potential. Treatment consists of PF00562271 tablets continued until progression of disease, unacceptable toxicity, or patient request. Evaluations for bioactivity are measured by serial FDG-PET and blood tests for biomarkers related to FAK and PYK2 kinase activities.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic, head and neck, and prostatic neoplasms, and patients with non-hematologic malignancies who have tumor appropriate for serial biopsy.
* Adequate organ function, including bilirubin less than 1.5 x ULN, and [Eastern Cooperative Oncology Group] ECOG performance status of 0-2.

Exclusion Criteria:

* Clinically significant gastrointestinal abnormalities, requirement for systemic anticoagulants or potent CYP 3A4 inhibitors, and history of clinically significant cardiac or pulmonary disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2005-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (2):
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Nashville, Tennessee
- Pfizer Investigational Site, East Melbourne, Victoria, Australia
- Pfizer Investigational Site, Toronto, Ontario, Canada

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8031001&StudyName=%20Study%20Of%20PF-00562271%2C%20Including%20Patients%20With%20Pancreatic%2C%20Head%20And%20Neck%2C%20Prostatic%20Neoplasms

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Expansion cohort (E1 or E2): participants were to be those enrolled at maximum tolerated dose level. E1: to have advanced disease likely to possess functional aberrations of pathways for tumorigenesis (represent focal adhesion kinase [FAK] expression). E2: to have disease characteristics associated with FAK expression and agree to repeat biopsies.
Groups:
- PF-00562271 5 mg BID: PF-00562271 administered as 5 milligrams (mg) orally (PO) twice a day (BID) without food (w/o food: no food within 2 hours prior to dosing) (escalation cohort).
- PF-00562271 10 mg BID: PF-00562271 administered as 10 mg PO BID w/o food (escalation cohort).
- PF-00562271 15 mg BID: PF-00562271 administered as 15 mg PO BID w/o food (escalation cohort).
- PF-00562271 25 mg BID: PF-00562271 administered as 25 mg PO BID w/o food (escalation cohort).
- PF-00562271 35 mg BID: PF-00562271 administered as 35 mg PO BID w/o food (escalation cohort).
- PF-00562271 45 mg BID: PF-00562271 administered as 45 mg PO BID w/o food (escalation cohort).
- PF-00562271 60 mg BID: PF-00562271 administered as 60 mg PO BID w/o food (escalation cohort).
- PF-00562271 75 mg BID: PF-00562271 administered as 75 mg PO BID with food (w/food: regular meal 200 to 800 calories) (expansion cohort).
  As of July 2008, participants newly enrolled to the expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration w/food): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3. Participant who was not able to titrate higher than 75 mg BID was reported in the 75 mg BID expansion cohort.
- PF-00562271 80 mg BID: PF-00562271 administered as 80 mg PO BID w/o food (escalation cohort).
- PF-00562271 100 mg BID: PF-00562271 administered as 100 mg BID w/food (escalation cohort). As of July 2008, participants newly enrolled to expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration w/food): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3. Participants who were not able to titrate higher than 100 mg BID were reported in the 100 mg BID cohort. Escalation and expansion cohorts were combined for reporting.
- PF-00562271 105 mg BID: PF-00562271 administered as 105 mg PO BID w/o food (escalation cohort).
- PF-00562271 125 mg BID: PF-00562271 administered as 125 mg PO BID w/food (escalation cohort). As of July 2008, participants newly enrolled to expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration w/food): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3.
  Additional participants were to be enrolled to the expansion cohort at the maximum tolerated dose (MTD) 125 mg BID (expansion cohort [E1 or E2]); E1 cohort United States (US) participants received Midazolam (MDZ) syrup 2 mg per milliliter (mg/mL) as a single PO dose 24 hours prior to first PF-00562271 dose (w/o food 2 hours prior to and after MDZ dosing) and on Cycle 1, Day 21 (C1.D21) simultaneously with PF-00562271 dosing (w/food). E1 participants outside the US and E2 participants were not dosed with MDZ.
  Escalation and expansion cohorts were combined for reporting.
- PF-00562271 150 mg BID: PF-00562271 administered as 150 mg PO BID w/food (escalation cohort).
- PF-00562271 125 mg QD: PF-00562271 administered as 125 mg PO once a day (QD) w/o food (escalation cohort).
- PF-00562271 175 mg QD: PF-00562271 administered as 175 mg PO QD w/o food (escalation cohort).
- PF-00562271 225 mg QD: PF-00562271 administered as 225 mg PO QD w/o food (escalation cohort).
Period: Overall Study
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 75 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Started | 2 | 4 | 3 | 4 | 3 | 4 | 4 | 1 | 3 | 10 | 6 | 33 | 3 | 4 | 7 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 4 | 3 | 4 | 3 | 4 | 4 | 1 | 3 | 10 | 6 | 33 | 3 | 4 | 7 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 0
Not completed — Laboratory abnormality | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 4 | 3 | 3 | 3 | 3 | 4 | 0 | 3 | 5 | 3 | 26 | 3 | 2 | 4 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 0 | 1 | 3 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: PF-00562271 dose escalation administered as 5 mg PO BID up to 150 mg PO BID or 125 mg PO QD up to 225 mg PO QD. Participants in the PF-00562271125 mg BID US E1 cohort administered MDZ 2 mg/mL as a single dose on C1.D1 and C1.D21 prior to PF-00562271 dosing.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 99
Age Continuous [Mean (Standard Deviation); unit: years] | 58.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Cycle Dose Limiting Toxicities (DLTs)
Description: At least possibly attributable to study treatment (Tx): Grade (Gr) 4 neutropenia (absolute neutrophil count [ANC] <500 cells/mm^3) for >7 days or Gr 3 febrile neutropenia (ANC <1000/mm^3, fever ≥38 degrees Celsius; Gr 4 thrombocytopenia (platelets <25,000 cells/mm^3); Gr ≥3 non-hematologic toxicity despite adequate medical intervention; Gr ≥3 confirmed prolonged QTc interval (>500 milliseconds [msec]); confirmed cardiac troponin I ≥99 percentile of reference range; Tx related toxicities with failure to receive ≥18 days Tx in 21-day cycle or inability to resume current dose level ≤14 days.
Time Frame: Baseline up to Cycle 1 Day 21 (C1.D21)
Population: Safety analysis set: All enrolled participants who started treatment.
Measure: Number; unit: participants
Groups:
- PF-00562271 75 mg BID: PF-00562271 administered as 75 mg PO BID with food (w/food: regular meal 200 to 800 calories) (escalation cohort).
  As of July 2008, participants newly enrolled to expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3. Participant who was not able to titrate higher than 75 mg BID was reported in the 75 mg BID cohort.
- PF-00562271 100 mg BID: PF-00562271 administered as 100 mg BID w/food (escalation cohort). As of July 2008, participants newly enrolled to expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3. Participants who were not able to titrate higher than 100 mg BID were reported in the 100 mg BID cohort.
- PF-00562271 125 mg BID: PF-00562271 administered as 125 mg PO BID w/food (escalation cohort). As of July 2008, participants newly enrolled to expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3.
  Additional participants were to be enrolled to the expansion cohort at the maximum tolerated dose (MTD) 125 mg BID (expansion cohort [E1 or E2]); E1 cohort United States (US) participants received Midazolam (MDZ) syrup 2 mg per milliliter (mg/mL) as a single PO dose 24 hours prior to first PF-00562271 dose (w/o food 2 hours prior to and after MDZ dosing) and on Cycle 1, Day 21 simultaneously with PF-00562271 dosing (w/food). E1 participants outside the US and E2 participants were not dosed with MDZ.
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 75 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 2 | 4 | 3 | 4 | 3 | 4 | 4 | 1 | 3 | 10 | 6 | 33 | 3 | 4 | 7 | 8
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1

2. Primary Outcome: Percentage of Participants With Tumor Metabolic Response (Reduction of ≥15%) in Positron Emission Tomography With F-18-fluorodeoxyglucose (FDG-PET)
Description: Metabolic response demonstrated in any tumor reduction of ≥15% in tumor FDG standardized uptake value (SUV) in Cycle 1; based on the recommendations of the European Organization for Research and Treatment of Cancer (EORTC) PET Study Group. Participant must have had a baseline PET with at least 1 tumor lesion demonstrating an FDG SUV of ≥5.
Time Frame: Baseline, C1.D14
Population: Participants in the 125 mg BID expansion cohort with at least 1 dose of study treatment, at least 1 lesion with an SUV ≥5 at baseline, and an on-study PET assessment C1.D14 (Day 13 up to Day 17).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- PF-00562271 125 mg BID: PF-00562271 administered as 125 mg PO BID w/food (escalation cohort). As of July 2008, participants newly enrolled to expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration w/food): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3.
  Additional participants were to be enrolled to the expansion cohort at the maximum tolerated dose (MTD) 125 mg BID (expansion cohort [E1 or E2]); E1 cohort United States (US) participants received Midazolam (MDZ) syrup 2 mg per milliliter (mg/mL) as a single PO dose 24 hours prior to first PF-00562271 dose (w/o food 2 hours prior to and after MDZ dosing) and on Cycle 1, Day 21 simultaneously with PF-00562271 dosing (w/food). E1 participants outside the US and E2 participants were not dosed with MDZ.
Arm/Group | PF-00562271 125 mg BID
Number analyzed (Participants) | 14
percentage of participants | 50 [26.4 to 73.6]

3. Secondary Outcome: Maximum Serum Concentration (Cmax): PF-00562271 C0.D1, C1.D1
Time Frame: Escalation cohorts: C0.D1 0 hour (0 hr=pre-dose PF-00562271), and 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hrs post dose; Expansion E1 US cohort: C1.D1 0 hr (prior to MDZ dose); E1 non-US and E2 cohort: C1.D1 0 hr and 0.5, 1, 2, 4 hrs post C1.D1 morning (am) dose
Population: Pharmacokinetic (PK) parameter analysis set: all participants with at least 1 dose of study treatment and at least 1 of the PK parameters of interest estimated in at least 1 treatment period. Escalation cohorts: Cycle 0 48 hours post dose timepoint = C1.D1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- PF-00562271 125 mg BID: PF-00562271 administered as 125 mg PO BID w/food (escalation cohort). As of July 2008, participants newly enrolled to expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3.
- PF-00562271 75 mg BID (Expansion Cohort): PF-00562271 administered as 75 mg PO BID with food w/food. As of July 2008, participants newly enrolled to the expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration w/food): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3. Participant who was not able to titrate higher than 75 mg BID was reported in the 75 mg BID expansion cohort.
- PF-00562271 100 mg BID (Expansion Cohort): PF-00562271 administered as 100 mg PO BID w/food. As of July 2008, participants newly enrolled to expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration w/food): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3. Participants who were not able to titrate higher than 100 mg BID were reported in the 100 mg BID cohort.
- PF-00562271 125 mg BID (Expansion Cohort): PF-00562271 administered as 125 mg PO BID w/food. As of July 2008, participants newly enrolled to expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration w/food): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3.
  Additional participants were to be enrolled to the expansion cohort at the maximum tolerated dose (MTD) 125 mg BID (expansion cohort [E1 or E2]); E1 cohort United States (US) participants received Midazolam (MDZ) syrup 2 mg per milliliter (mg/mL) as a single PO dose 24 hours prior to first PF-00562271 dose (w/o food 2 hours prior to and after MDZ dosing) and on Cycle 1, Day 21 simultaneously with PF-00562271 dosing (w/food). E1 participants outside the US and E2 participants were not dosed with MDZ.
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD | PF-00562271 75 mg BID (Expansion Cohort) | PF-00562271 100 mg BID (Expansion Cohort) | PF-00562271 125 mg BID (Expansion Cohort)
Number analyzed (Participants) | 2 | 4 | 3 | 4 | 3 | 4 | 4 | 3 | 3 | 6 | 7 | 3 | 4 | 7 | 8 | 1 | 4 | 11
nanograms per milliliter (ng/mL) | 49.63 (4) | 71.13 (24) | 138.8 (73) | 130.1 (176) | 306.1 (28) | 312.9 (108) | 363.2 (37) | 597.6 (2) | 397.3 (91) | 1018 (48) | 1236 (49) | 647.2 (52) | 1110 (35) | 1528 (57) | 2605 (35) | 421.0 (0) | 474.6 (44) | 747.9 (75)

4. Secondary Outcome: Maximum Serum Concentration (Cmax): PF-00562271 C1.D14
Time Frame: Escalation and Expansion E1 and E2 cohorts: C1.D14 0 hour (0 hr=pre-dose PF-00562271), and 0.5, 1, 2, 4, 6, 8, 12 (if BID) or 24 (if QD) hrs post am dose
Population: PK parameter analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 2 | 4 | 3 | 4 | 3 | 3 | 4 | 3 | 4 | 4 | 7 | 2 | 4 | 5 | 4
ng/mL | 74.65 (80) | 134.7 (55) | 309.6 (58) | 307.7 (145) | 655.4 (72) | 1105 (46) | 1083 (84) | 1767 (61) | 2295 (74) | 2580 (62) | 2947 (62) | 3445 (65) | 2021 (17) | 3136 (43) | 4438 (49)

5. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax): PF-00562271 C0.D1, C1.D1
Time Frame: Escalation cohorts: C0.D1 0 hour (0 hr=pre-dose PF-00562271), and 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hrs post dose; Expansion E1 US cohort: C1.D1 0 hr (prior to MDZ dose); E1 non-US and E2 cohort: C1.D1 0 hr and 0.5, 1, 2, 4 hrs post C1.D1 am dose
Population: PK parameter analysis set. Escalation cohorts: Cycle 0 48 hours post dose timepoint = C1.D1.
Measure: Median (Full Range); unit: hours
Groups:
- PF-00562271 100 mg BID: PF-00562271 administered as 100 mg BID w/food (escalation cohort). As of July 2008, participants newly enrolled to the expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3. Participants who were not able to titrate higher than 100 mg BID were reported in the 100 mg BID cohort.
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD | PF-00562271 75 mg BID (Expansion Cohort) | PF-00562271 100 mg BID (Expansion Cohort) | PF-00562271 125 mg BID (Expansion Cohort)
Number analyzed (Participants) | 2 | 4 | 3 | 4 | 3 | 4 | 4 | 3 | 3 | 6 | 7 | 3 | 4 | 7 | 8 | 1 | 4 | 11
hours | 0.500 [0.500 to 0.500] | 1.50 [1.00 to 2.00] | 0.500 [0.500 to 1.00] | 0.500 [0.500 to 0.500] | 1.00 [0.500 to 2.00] | 1.50 [1.00 to 4.00] | 1.00 [1.00 to 2.00] | 2.00 [0.500 to 8.00] | 4.00 [4.00 to 4.00] | 2.00 [0.500 to 6.00] | 4.00 [0.500 to 8.00] | 4.00 [0.500 to 8.00] | 5.00 [4.00 to 6.00] | 4.00 [2.00 to 6.00] | 4.00 [2.00 to 6.00] | 4.00 [4.00 to 4.00] | 6.00 [4.00 to 8.00] | 4.00 [1.00 to 4.00]

6. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax): PF-00562271 C1.D14
Time Frame: as for outcome 4
Population: PK parameter analysis set
Measure: Median (Full Range); unit: hours
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 2 | 4 | 3 | 4 | 3 | 3 | 4 | 3 | 4 | 4 | 7 | 2 | 4 | 5 | 4
hours | 0.500 [0.500 to 0.500] | 1.00 [0.500 to 2.00] | 1.00 [1.00 to 8.00] | 1.50 [0.500 to 4.00] | 2.00 [2.00 to 12.0] | 1.00 [0.500 to 4.00] | 1.50 [1.00 to 4.00] | 2.00 [1.00 to 2.00] | 2.25 [0.000 to 12.0] | 3.00 [0.500 to 4.00] | 4.00 [0.000 to 12.0] | 7.00 [6.00 to 8.00] | 5.00 [2.00 to 8.00] | 2.00 [2.00 to 4.00] | 2.50 [0.500 to 8.00]

7. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast): PF-00562271 C0.D1, C1.D1
Description: Area under the serum concentration time-curve from zero to the last measured concentration; nanograms multiplied by hours per milliliters (ng*hr/mL).
Time Frame: as for outcome 5
Population: PK parameter analysis set. Escalation cohorts: Cycle 0 48 hours post dose timepoint = C1.D1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 2 | 4 | 3 | 4 | 3 | 4 | 4 | 3 | 3 | 6 | 7 | 3 | 4 | 7 | 8
ng*hr/mL | 81.13 (47) | 233.8 (14) | 348.1 (67) | 295.6 (213) | 1205 (6) | 2364 (118) | 1735 (67) | 4407 (42) | 3501 (171) | 10600 (61) | 11900 (163) | 6083 (134) | 16330 (12) | 20830 (66) | 38600 (78)

8. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf): PF-00562271 C0.D1, C1.D1
Description: AUCinf = area under the serum concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: as for outcome 5
Population: PK parameter analysis set. Escalation cohorts: Cycle 0 48 hours post dose timepoint = C1.D1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 3 | 4 | 4 | 3 | 2 | 5 | 3 | 3 | 4 | 7 | 6
ng*hr/mL | 86.24 (48) | 239.6 (14) | 354.1 (68) | 574.1 (18) | 1222 (6) | 2399 (118) | 1759 (66) | 4507 (44) | 6588 (65) | 10880 (71) | 5534 (271) | 6101 (135) | 16770 (13) | 21190 (65) | 37560 (87)

9. Secondary Outcome: Serum Decay Half-life (t 1/2): PF-00562271 C0.D1, C1.D1
Description: Serum decay half-life is the time measured for the serum concentration to decrease by one half.
Time Frame: as for outcome 5
Population: PK parameter analysis set. Escalation cohorts: Cycle 0 48 hours post dose timepoint = C1.D1.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 3 | 4 | 4 | 3 | 2 | 5 | 3 | 3 | 4 | 7 | 6
hours | 1.990 (0.60811) | 2.078 (0.40901) | 2.173 (0.38799) | 2.837 (1.2176) | 2.897 (0.53304) | 5.270 (1.8993) | 3.365 (0.88410) | 4.770 (0.51069) | 5.025 (0.62933) | 6.180 (2.9592) | 3.853 (1.4332) | 4.407 (1.9318) | 8.388 (1.9370) | 5.937 (1.1016) | 7.948 (2.7254)

10. Secondary Outcome: Apparent Oral Clearance (CL/F): PF-00562271 C0. D1, C1.D1
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: as for outcome 5
Population: PK parameter analysis set. Escalation cohorts: Cycle 0 48 hours post dose timepoint = C1.D1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per minute (mL/min)
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 2 | 5 | 3 | 3 | 4 | 7 | 6
milliliters per minute (mL/min) | 964.2 (48) | 702.1 (17) | 707.2 (68) | 726.0 (18) | 478.0 (6) | 312.3 (118) | 568.3 (66) | 295.5 (44) | 253.2 (64) | 160.9 (71) | 475.5 (553) | 516.9 (120) | 124.0 (13) | 137.7 (65) | 99.85 (87)

11. Secondary Outcome: Minimum Observed Serum Trough Concentration (Cmin): PF-00562271 C1.D14
Time Frame: as for outcome 4
Population: PK parameter analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 2 | 4 | 3 | 4 | 3 | 3 | 4 | 3 | 4 | 4 | 7 | 2 | 4 | 5 | 4
ng/mL | 0.01349 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 0.8059 (12668339981) | 48.96 (89) | 33.11 (1046) | 145.8 (131) | 315.3 (112) | 359.8 (80) | 594.5 (134) | 1005 (117) | 1131 (67) | 1253 (86) | 0.4111 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 439.6 (48) | 634.7 (92) | 1129 (123)

12. Secondary Outcome: Area Under the Curve From Time Zero to the End of the Dosing Interval (AUCtau): PF-00562271 C1.D14
Time Frame: as for outcome 4
Population: PK parameter analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 2 | 4 | 3 | 4 | 3 | 3 | 4 | 3 | 4 | 4 | 7 | 2 | 4 | 5 | 2
ng*hr/mL | 156.3 (53) | 447.2 (122) | 1573 (80) | 1476 (238) | 4519 (84) | 8357 (61) | 8173 (74) | 12920 (86) | 20010 (76) | 21120 (62) | 24340 (77) | 26200 (22) | 24470 (30) | 43140 (50) | 68780 (71)

13. Secondary Outcome: Observed Accumulation Ratio (Rac): PF-00562271 C1.D14
Description: Rac was the ratio of the Day 14 AUC0-tau (0 hour to last dose interval) and AUC during the corresponding time period after the lead-in dose (AUCtau C1.D14/AUCtau C0.D1).
Time Frame: Escalation (Esc) cohort: C0.D1: 0 hr, and 0.5, 1, 2, 4, 6, 7,12 hrs post dose; Expansion (Exp) cohort: C0:D1: 0 hr, and 1, 2, 4, 8 hrs post dose; Esc and Exp cohorts: C1.D14 0 hour, and 0.5, 1, 2, 4, 6, 8, 12 (if BID) or 24 (if QD) hrs post am dose
Population: PK parameter analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 2 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 3 | 4 | 5 | 3 | 5 | 2
ratio | 1.864 (4) | 2.997 (26) | 4.522 (50) | 5.061 (66) | 3.899 (80) | 5.038 (125) | 5.060 (99) | 3.638 (45) | 5.581 (57) | 2.967 (18) | 3.608 (49) | 1.961 (20) | 2.293 (52) | 1.118 (60)

14. Secondary Outcome: Maximum Serum Concentration (Cmax): MDZ
Time Frame: C0.D1, C1.D21 Expansion cohort E1 US sites only: 0 hr (prior to MDZ dosing) and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hrs post MDZ dose
Population: N=participants in the PK parameter analysis set who received MDZ dosing prior to PF-00562271 in the 125 mg BID cohort; (n)=number of participants with analyzable data at observation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-00562271 125 mg BID
Number analyzed (Participants) | 11
ng/mL
  C0.D1 (n=11) | 13.14 (47)
  C1.D21 (n=8) | 20.40 (31)
Statistical Analysis 1: Comparison: PF-00562271 125 mg BID; Participants in the PF-00562271 125 mg BID cohort who received MDZ (test) administered prior to PF-00562271 (reference) dosing; Test type: Superiority or Other; Ratio (percent) test / reference = 155.66, 90% CI 2-sided [109.66 to 220.95] — Ratio of adjusted geometric means Day 21 versus Day 1. Values have been transformed from the log scale

15. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast): MDZ
Description: Area under the serum concentration time-curve from zero to the last measured concentration.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-00562271 125 mg BID
Number analyzed (Participants) | 11
ng*hr/mL
  C0.D1 (n=11) | 42.44 (53)
  C1.D21 (n=8) | 134.0 (22)
Statistical Analysis 1: Comparison: PF-00562271 125 mg BID; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; Ratio (percent) test / reference = 315.72, 90% CI 2-sided [227.60 to 437.97] — Ratio of adjusted geometric means Day 21 versus Day 1. Values have been transformed from the log scale

16. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf): MDZ
Description: as for outcome 8
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-00562271 125 mg BID
Number analyzed (Participants) | 11
ng*hr/mL
  C0.D1 (n=11) | 49.79 (61)
  C1.D21 (n=5) | 212.3 (24)
Statistical Analysis 1: Comparison: PF-00562271 125 mg BID; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; Ratio (percent) test / reference = 496.63, 90% CI 2-sided [206.24 to 1195.92] — Ratio of adjusted geometric means Day 21 versus Day 1. Values have been transformed from the log scale

17. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax): MDZ
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | PF-00562271 125 mg BID
Number analyzed (Participants) | 11
hours
  C0.D1 (n=11) | 0.500 [0.500 to 1.00]
  C1.D21 (n=8) | 1.00 [0.500 to 3.00]

18. Secondary Outcome: Serum Decay Half-life (t 1/2): MDZ
Description: Serum decay half-life is the time measured for the serum concentration to decrease by one half.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-00562271 125 mg BID
Number analyzed (Participants) | 11
hours
  C0.D1 (n=11) | 5.045 (1.7221)
  C1.D21 (n=5) | 7.764 (0.68475)

19. Secondary Outcome: Apparent Oral Clearance (CL/F): MDZ
Description: as for outcome 10
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | PF-00562271 125 mg BID
Number analyzed (Participants) | 11
mL/hr
  C0.D1 (n=11) | 20090 (61)
  C1.D21 (n=5) | 4709 (24)

20. Secondary Outcome: Percentage of Participants With Best Overall Response as Measured Using the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Best response recorded from start of treatment (Tx) until disease progression. Complete response: disappearance of all target lesions. Partial response: ≥30% decrease in sum of longest dimensions (LD) of target lesions referencing baseline sum LD. Progressive disease: ≥20% increase in sum LD of target lesions from smallest sum LD recorded since Tx start or appearance of ≥1 new lesions. Stable disease: neither sufficient shrinkage to=PR nor sufficient increase to=PD during first 6 weeks after Tx start referencing smallest sum LD since Tx start.
Time Frame: Baseline up to 12 cycles (cycle=21days)
Population: RECIST response analysis set: all enrolled participants who had an adequate baseline tumor assessment, measureable disease and who started treatment. N=number of participants with evaluable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 75 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 2 | 4 | 3 | 4 | 3 | 2 | 4 | 1 | 3 | 8 | 6 | 31 | 3 | 3 | 6 | 8
percentage of participants
  Complete response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable disease | 0 | 1 | 2 | 2 | 2 | 0 | 2 | 0 | 2 | 2 | 2 | 11 | 0 | 1 | 3 | 1
  Progressive disease | 2 | 3 | 1 | 2 | 1 | 1 | 2 | 0 | 1 | 2 | 4 | 15 | 3 | 2 | 2 | 3
  Indeterminate | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 5 | 0 | 0 | 1 | 4

21. Secondary Outcome: Phosphorylated Focal Adhesion Kinase (pFAK)
Description: Analysis of tumor specimens to assess FAK-related biomarkers for potential predictors of response markers to PF-00562271; FAK is overexpressed in a variety of human cancers. For dose escalation cohorts and expansion cohort E1, pre-treatment tumor biopsy collected between Day -28 and first PF-00562271 dose and on-treatment tumor biopsy collected 2 to 8 hours after PF-00562271 dose during Cycle 1 between day 12 and 16. In addition, up to 10 participants in cohort E2 were to be enrolled for serial biopsies.
Time Frame: Baseline (up to 28 days prior to first dose) up to 12 cycles (cycle=21days)
Population: Data was not summarized as samples were processed and analyzed later than 3 days after collection and thus the data were considered unusable.
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 75 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Phosphorylated Mitogen Activated Pathway Kinase (pMAPK)
Description: Analysis of tumor specimens to assess FAK-related biomarkers for potential predictors of response markers to PF-00562271; MAPK regulates activities of several transcription factors. A defect in MAPK pathway leads to uncontrolled cell growth. For dose escalation cohorts and expansion cohort E1, pre-treatment tumor biopsy collected between Day -28 and first PF-00562271 dose and on-treatment tumor biopsy collected 2 to 8 hours after PF-00562271 dose during Cycle 1 between day 12 and 16. In addition, up to 10 participants in cohort E2 were to be enrolled for serial biopsies.
Time Frame: Baseline (up to 28 days prior to first dose) up to 12 cycles (cycle=21days)
Population: as for outcome 21
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 75 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Phospho-SRC (pSRC)
Description: Analysis of tumor specimens to assess FAK-related biomarkers for potential predictors of response markers to PF-00562271; SRC proto-oncogenes are regulators of growth and differentiation of eukaryotic cells and are implicated in development of human tumors. For dose escalation cohorts and expansion cohort E1, pre-treatment tumor biopsy collected between Day -28 and first PF-00562271 dose; on-treatment tumor biopsy collected 2 to 8 hours after PF-00562271 dose during Cycle 1 between day 12 and 16. In addition, up to 10 participants in cohort E2 were to be enrolled for serial biopsies.
Time Frame: Baseline (up to 28 days prior to first dose) up to 12 cycles (cycle=21days)
Population: as for outcome 21
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 75 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Caspase-3
Description: Analysis of tumor specimens to assess FAK-related biomarkers for potential predictors of response markers to PF-00562271; sequential activation of caspases plays a central role in the execution-phase of cell apoptosis. For dose escalation cohorts and expansion cohort E1, pre-treatment tumor biopsy collected between Day -28 and first PF-00562271 dose and on-treatment tumor biopsy collected 2 to 8 hours after PF-00562271 dose during Cycle 1 between day 12 and 16. In addition, up to 10 participants in cohort E2 were to be enrolled for serial biopsies.
Time Frame: Baseline (up to 28 days prior to first dose) up to 12 cycles (cycle=21days)
Population: as for outcome 21
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 75 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are recorded from the time of first dose of study treatment up to 28 days after last dose of study treatment or until start of new anti-cancer treatment, whichever occurs first.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- PF-00562271 125 mg BID: PF-00562271 administered as 125 mg PO BID w/food (escalation cohort). As of July 2008, participants newly enrolled to expansion cohort or who restarted treatment after dose delay associated with adverse event(s) were dosed according to intra-participant escalation (up-titration w/food): 75 mg BID week 1; 100 mg BID week 2; 125 mg BID week 3.
  Additional participants were to be enrolled to the expansion cohort at the maximum tolerated dose (MTD) 125 mg BID (expansion cohort [E1 or E2]); E1 cohort United States (US) participants received Midazolam (MDZ) syrup 2 mg per milliliter (mg/mL) as a single PO dose 24 hours prior to first PF-00562271 dose (w/o food 2 hours prior to and after MDZ dosing) and on Cycle 1, Day 21 simultaneously with PF-00562271 dosing (w/food). E1 participants outside the US and E2 participants were not dosed with MDZ.
  Escalation and expansion cohorts were combined for reporting.
Arm/Group | PF-00562271 5 mg BID | PF-00562271 10 mg BID | PF-00562271 15 mg BID | PF-00562271 25 mg BID | PF-00562271 35 mg BID | PF-00562271 45 mg BID | PF-00562271 60 mg BID | PF-00562271 75 mg BID | PF-00562271 80 mg BID | PF-00562271 100 mg BID | PF-00562271 105 mg BID | PF-00562271 125 mg BID | PF-00562271 150 mg BID | PF-00562271 125 mg QD | PF-00562271 175 mg QD | PF-00562271 225 mg QD
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/4 | 0/3 | 0/4 | 2/3 | 1/4 | 2/4 | 0/1 | 0/3 | 3/10 | 3/6 | 12/33 | 0/3 | 0/4 | 0/7 | 3/8
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 3/3 | 4/4 | 3/3 | 4/4 | 4/4 | 1/1 | 3/3 | 10/10 | 6/6 | 33/33 | 3/3 | 4/4 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00562271 5 mg BID (N=2) | PF-00562271 10 mg BID (N=4) | PF-00562271 15 mg BID (N=3) | PF-00562271 25 mg BID (N=4) | PF-00562271 35 mg BID (N=3) | PF-00562271 45 mg BID (N=4) | PF-00562271 60 mg BID (N=4) | PF-00562271 75 mg BID (N=1) | PF-00562271 80 mg BID (N=3) | PF-00562271 100 mg BID (N=10) | PF-00562271 105 mg BID (N=6) | PF-00562271 125 mg BID (N=33) | PF-00562271 150 mg BID (N=3) | PF-00562271 125 mg QD (N=4) | PF-00562271 175 mg QD (N=7) | PF-00562271 225 mg QD (N=8)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureteral disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00562271 5 mg BID (N=2) | PF-00562271 10 mg BID (N=4) | PF-00562271 15 mg BID (N=3) | PF-00562271 25 mg BID (N=4) | PF-00562271 35 mg BID (N=3) | PF-00562271 45 mg BID (N=4) | PF-00562271 60 mg BID (N=4) | PF-00562271 75 mg BID (N=1) | PF-00562271 80 mg BID (N=3) | PF-00562271 100 mg BID (N=10) | PF-00562271 105 mg BID (N=6) | PF-00562271 125 mg BID (N=33) | PF-00562271 150 mg BID (N=3) | PF-00562271 125 mg QD (N=4) | PF-00562271 175 mg QD (N=7) | PF-00562271 225 mg QD (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dysacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endocrine disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 4 | 1 | 0 | 1 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 6 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 1 | 2 | 1 | 0 | 0 | 4 | 4 | 10 | 2 | 2 | 4 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 3 | 2 | 1 | 3 | 4 | 3 | 22 | 2 | 4 | 7 | 8
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 1 | 3 | 6 | 3 | 15 | 3 | 3 | 4 | 7
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 4 | 1 | 2 | 1 | 1 | 1 | 3 | 3 | 16 | 1 | 4 | 3 | 6
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 4 | 3 | 12 | 0 | 0 | 3 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 3 | 1 | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood prolactin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 2 | 9 | 0 | 0 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 8 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 2 | 6 | 2 | 2 | 3 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 4 | 3 | 14 | 3 | 2 | 6 | 4
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 5 | 1 | 2 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 2 | 6 | 0 | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Corrective lens user (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 8 | 1 | 0 | 0 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
PET and RECIST Response Analysis Sets as defined in Protocol Amendment 3 dated 20Mar2007 are reported in Basic Results per the revised definitions in Statistical Analysis Plan version 2 dated 11Apr2008.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.